CLINICAL TRIAL: NCT00309387
Title: Collaborative Italian-American Clinical Trial of Nutritional Supplements and Age-related Cataract (CTNS)
Acronym: CTNS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEI-110
Record Dates: First submitted 2006-03-29; First posted 2006-03-31 (Estimated); Results first posted 2012-04-24 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-04

CONDITIONS: Cataract
Keywords: Cataract; Nutritional supplements
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Centrum (Experimental): multivitamin-mineral supplement. RDA dosage. 1 tablet a day for the whole study duration.
  Interventions: Dietary Supplement: Centrum
- placebo (Placebo Comparator): placebo pills. One tablet a day for the whole study duration.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Centrum — Multivitamin/mineral supplement containing US RDA levels of nutrients. 1 tablet a day for the expected duration of follow-up (on average 10 yrs).
  Arms: Centrum
Other: Placebo — placebo tablets manufactured to mimic Centrum tablets.
  Arms: placebo

SUMMARY:
The Collaborative Italian-American Clinical Trial of Nutritional Supplements and Age-related Cataract (CTNS) is a 13-year study designed primarily to evaluate the safety and efficacy of a vitamin-mineral supplement (Centrum) containing recommended daily-allowance dosage (RDA) in preventing age-related cataract or delaying its progression in participants with early or no cataract at baseline.

DETAILED DESCRIPTION:
Despite dramatic increase in the rates of cataract surgery during the last decades, age-related cataract is still responsible for about 50% of cases of severe visual impairment in developing countries, and for high and growing health care costs in western countries. CTNS was designed to complement the U.S. Age-Related Eye Disease Study (AREDS) by evaluating a much broader spectrum of nutrients at RDA dosages. Whereas about 60% of the AREDS control group was taking RDA dose multivitamin supplements, none of the participants in CTNS had taken any type of nutritional supplement for at least one year before the qualification visit. Therefore, the CTNS will be able to evaluate the effect of RDA doses versus no supplementation at all. CTNS and AREDS will use similar procedures, including those for grading the presence and severity of lens changes.

CTNS is a randomized,parallel group, placebo controlled, double blinded, single center, intervention trial.

Primary Outcomes: photographic evaluation of a prespecified increase from baseline in nuclear, cortical, or posterior subcapsular cataract (PSC) opacity grades or cataract surgery.

Secondary Outcomes: increase in type-specific opacity grade, cataract surgery, and visual acuity loss from baseline > or = 15 letters.

Patients will be followed for a maximum of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and photographic diagnosis of early or no age-related cataract
* Participants with early cataract must have at least one eligible eye with VA score 20/32 or better
* Participants with no cataract must have VA score 20/32 or better in both eyes.

Exclusion Criteria:

* Advanced cataract
* Bilateral aphakia or pseudophakia
* Any ocular disease or condition that might complicate the future evaluation of cataract
* Regular use of nutritional supplements
* Failure to take at least 75% of run-in medication
* Cancer with evidence of recurrence in the past 5 years
* Major cerebral or cardiovascular events in past 12 months
* Current participation to other clinical trials
* Any condition likely to prevent adherence to CTNS follow-up schedule

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 1995-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Maraini, MD, Study Chair — University of Parma; Robert D Sperduto, MD, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- Dpt. Scienze Otorino-Odonto Oftalmologiche, University of Parma, Parma, Italy

REFERENCES:
- [Background] CTNS Study Group. The Italian-American Clinical Trial of Nutritional Supplements and Age-Related Cataract (CTNS): design implications. CTNS report no. 1. Control Clin Trials. 2003 Dec;24(6):815-29. doi: 10.1016/s0197-2456(03)00095-3. PMID 14662284
- [Result] Ferrigno L, Aldigeri R, Rosmini F, Sperduto RD, Maraini G; Italian-American Cataract Study Group. Associations between plasma levels of vitamins and cataract in the Italian-American Clinical Trial of Nutritional Supplements and Age-Related Cataract (CTNS): CTNS Report #2. Ophthalmic Epidemiol. 2005 Apr;12(2):71-80. doi: 10.1080/09286580590932815. PMID 16019690
- [Result] Clinical Trial of Nutritional Supplements and Age-Related Cataract Study Group; Maraini G, Williams SL, Sperduto RD, Ferris F, Milton RC, Clemons TE, Rosmini F, Ferrigno L. A randomized, double-masked, placebo-controlled clinical trial of multivitamin supplementation for age-related lens opacities. Clinical trial of nutritional supplements and age-related cataract report no. 3. Ophthalmology. 2008 Apr;115(4):599-607.e1. doi: 10.1016/j.ophtha.2008.01.005. PMID 18387406
- [Result] Maraini G, Williams SL, Sperduto RD, Ferris FL, Milton RC, Clemons TE, Rosmini F, Ferrigno L. Effects of multivitamin/mineral supplementation on plasma levels of nutrients. Report No. 4 of the Italian-American clinical trial of nutritional supplements and age-related cataract. Ann Ist Super Sanita. 2009;45(2):119-27. PMID 19636163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1020 participants were enrolled from January 8, 1996 through April 10, 1998 at the Institute of Ophthalmology of the University of Parma, Parma, Italy
Pre-assignment Details: Potential participants had to complete a 1-month placebo run-in period (use of > 75% of the run-in tablets) before randomization
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 510 | 510
Completed | 368 | 351
Not Completed | 142 | 159
Not completed — Death | 72 | 73
Not completed — Lost to Follow-up | 70 | 86

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 510 | 510 | 1020
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 139 | 140 | 279
  >=65 years | 371 | 370 | 741
Age Continuous [Mean (Standard Deviation); unit: years] | 67.7 (4.82) | 67.7 (4.97) | 67.7 (4.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 226 | 459
  Male | 277 | 284 | 561
Region of Enrollment [Number; unit: participants]
  Italy | 510 | 510 | 1020

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Showing Development or Progression of Age-related Cataract or Undergoing Cataract Surgery During Follow-up
Description: number of participants in whom any of the following occur in at least one eligible eye during follow-up: cataract surgery; nuclear opacity: a 1.5 U increase in opalescence from baseline; cortical opacity: a 10% increase in area within a standard 5 mm circle area of the lens from baseline; posterior subcapsular opacity: a 5% increase in area within a standard 5 mm circle area of the lens from baseline.
Time Frame: at yearly intervals from baseline for approximately ten years
Population: Intention to treat analysis
Measure: Number; unit: participants
Groups:
- Treatment: Centrum
- Placebo: Placebo
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 510 | 510
participants | 227 | 255
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.03, Regression, Cox; Cox Proportional Hazard = 0.82, 95% CI 2-sided [0.68 to 0.98]

2. Secondary Outcome: Number of Participants Showing Development or Progression of Nuclear Lens Opacities
Description: number of participants with a 1.5 U increase in nuclear opalescence from baseline in at least one eligible eye during follow-up
Time Frame: at yearly intervals from baseline for approximately ten years
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 510 | 510
participants | 84 | 118

3. Secondary Outcome: Number of Participants Showing Development or Progression of Cortical Lens Opacities
Description: Number of participants with a 10% increase in area of cortical opacity within a standard central 5 mm circle of the lens from baseline in at least one eligible eye during follow-up
Time Frame: at yearly intervals from baseline for approximately ten years
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 510 | 510
participants | 96 | 118

4. Secondary Outcome: Number of Participants Showing Development or Progression of Posterior Subcapsular Opacities
Description: Number of participants with a 5% increase in area of posterior subcapsular opacity within a standard central 5 mm circle of the lens from baseline in at least one eligible eye during follow-up
Time Frame: at yearly intervals from baseline for approximately ten years
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 510 | 510
participants | 74 | 37

5. Secondary Outcome: Number of Participants Undergoing Cataract Surgery
Description: number of participants undergoing cataract surgery in at least one eligible eye during follow-up
Time Frame: at 6 month intervals from baseline for approximately 10 yrs
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 510 | 510
participants | 88 | 90

6. Secondary Outcome: Number of Participants With a Decrease in Visual Acuity
Description: Number of participants with a decrease in best corrected visual acuity score from baseline of > 15 letters in at least one eligible eye during follow-up
Time Frame: at 6 month intervals from baseline for approximately 10 yrs
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 510 | 510
participants | 144 | 139

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 363/510 | 397/510
Other Adverse Events (participants affected / at risk) | 39/510 | 38/510
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=510) | Placebo (N=510)
death (General disorders) | 77 | 81
hospitalization (General disorders) | 286 (573) | 316 (604)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=510) | Placebo (N=510)
upset stomach (Gastrointestinal disorders) | 17 (17) | 19 (19)
increased weight (General disorders) | 3 (3) | 3 (3)
skin rash (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
other (General disorders) | 14 (14) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No